CLINICAL TRIAL: NCT05431829
Title: Analysis of Psychometric Properties and Cultural Adaptation of Urdu Version of Fonseca Anamnestic Index in Pakistani Population
Brief Title: Urdu Version of Fonseca Anamnestic Index: Reliability and Validity Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00255
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Temporomandibular Disorder
Keywords: Fonseca Anamnestic Index; Urdu Version; Reliability; Validity; Temporomandibular Disorder; General Population
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of study is to translate and culturally adapt Fonseca Anamnestic Index into Urdu language and to investigate the reliability and validity in Pakistani population over the age 18 years.

DETAILED DESCRIPTION:
The English version of the Fonseca Anamnestic Index will be translated and culturally adapted as per previous recommendation. In Pakistani general population, Urdu Version of Fonseca Anamnestic Index will distributed among 140 participants choose by random sampling technique based on pre-defined inclusion and exclusion criteria. To test inter and intra-observer reliability of the final Urdu Version of Fonseca Anamnestic Index questionnaire will be filled on the same day, by two observers, and for the Inter-Observers assessment, with an interval of 30 minute between the first and the second application. Third assessment will carried out after 7 days by Observer-1, for intra-observer assessment. Data will be entered and analyzed using Statistical Package of Social Sciences Version 24. Internal consistency will be analyzed with Cronbach alpha value. Test- re-test reliability will be assessed using an intra-class correlation coefficient. The Urdu Version of Fonseca Anamnestic Index will be evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient with the age of 18 years.
* Having any previous history of temporo-mandibular joint pain
* Having any current condition of temporo-mandibular disorders.
* Both Genders are included equally.

Exclusion Criteria:

* Inability to understand or follow the instructions of the Fonseca Anamnestic Index.
* Suffering from any neurological condition.
* Suffering from any unstable medical condition.
* Patients with rheumatoid arthritis were also excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani population with or without temporo-mandibular disorders over the age 18-80 years and both genders.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-10 (Estimated); Study Completion 2022-07-12 (Estimated)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index | 1st day
  It is a scale proposed to identify and determine the severity of temporo-mandibular disorder through 10 question being designed in the form of a questionnaire which is then to be filled and completed by the population.
Numeric Pain Rating Scale | 1st day
  The numeric pain rating scale is a self-implemented pain intensity perception scale. In this test, all the possibilities are arranged at the same level, with 0 being the absence of pain and 10 being the maximum pain
Short Form - 36 | 1st day
  The Short Form - 36 which is self-administered and evaluates general quality of life from physical and emotional points of view. It consists of 12 questions that are presented with a variable number of answers.
Dizziness Handicap Inventory | 1st day
  Dizziness and vertigo sensations were measured with the dizziness handicap inventory, which is a self-implemented scale that identifies vertigo or lack of balance. The instrument consists of 25 questions that can be answered as yes, no or sometimes. This questionnaire identifies functional, physical and emotional problems related to balance disorders.
Headache impact Test-6 | 1st day
  The headache impact test is a self-administered headache questionnaire that consists of six questions with five possible answers. The possible outcomes are "never", "rarely", "sometimes", "very often" and "always". The numerical result is the sum of the answers.
Neck Disability Index | 1st day
  The neck disability index is a questionnaire that assesses disability produced by neck pain. It consists of ten questions with six different answers that are ordered from least to most disability, with 0 corresponding to no disability and 5 corresponding to greatest disability. The result is the sum of the answers, ranging from 0 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No